CLINICAL TRIAL: NCT03521336
Title: The Effect of Intrathecal Transplantation of Umbilical Cord Mesenchymal Stem Cells in Patients With Sub-Acute Spinal Cord Injury：A Multicenter, Randomized, Controlled Trial
Brief Title: Intrathecal Transplantation of UC-MSC in Patients With Sub-Acute Spinal Cord Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: West China Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Limin Rong, Professor, President, Director of Department of Spine Surgery, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IT-UCMSC-SASCI
Record Dates: First submitted 2018-04-12; First posted 2018-05-11 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Umbilical Cord Mesenchymal Stem Cells
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: A 2:1 ratio of randomization (intervention group:control group) was used.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Mesenchymal Stem Cells (Experimental): Intrathecal Transplantation of Umbilical Cord Mesenchymal Stem Cells, 1*10^6 cells/kg, once a month for 4 months
  Interventions: Drug: Umbilical Cord Mesenchymal Stem Cells
- Control (Placebo Comparator): Placebo: Sham operation, 10ml saline, once a month for 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Umbilical Cord Mesenchymal Stem Cells — Intrathecal Transplantation of Umbilical Cord Mesenchymal Stem Cells
  Other Names: UC-MSC
  Arms: Umbilical Cord Mesenchymal Stem Cells
Drug: Placebo — Saline，Sham operation
  Other Names: Sham operation
  Arms: Control

SUMMARY:
This study aim to evaluate the safety and efficacy of intrathecal transplantation of allogeneic umbilical cord derived mesenchymal stem cells (UC-MSC) for treatment of different phrases of spinal cord injury. Here, the history of spinal cord injury is divided into three periods, Sub-acute SCI, Early stage of chronic SCI, and Late stage of chronic SCI, which is 2W-2M, 2M-12M, and more than 12M after injury, respectively. The purpose is to investigate whether the patients with spinal cord injury benefit from UC-MSC transplantation, and then find out the best time for SCI treatment.

In this part of the study, the investigators will treat patients with sub-acute spinal cord injury with UC-MSC transplantation or placebo.

DETAILED DESCRIPTION:
Spinal cord injury (SCI), damage to any part of the spinal cord or nerves, often causes permanent neurofunction deficit, including strength, sensation and other body functions below the site of injury. WHO reported 15-40/million people suffer from SCI each year, about 250,000 to 500,000 people. The majority of SCI victims are young patients, who are at the time of working age. As a result of that, SCI not only affects the physical and psychological health of those patients, but also bring huge economic burden to their families, as well as the society. The current treatments for SCI mainly include surgical operation, neuroregenerative medicine, physical therapy, chinese acupuncture and so on. However, none of these methods are efficient enough to make any functional recovery of neurological injury in patients, and most patients will have to face paraplegia or tetraplegia.

The most challenge of SCI treatment are reported to be regeneration of axon and rewiring of the damaged spinal cord. The properties of strong proliferation and differentiation make stem cell transplantation possible to replace the damage axon and rebridge the injury spinal cord. Currently, evidences from animal experiments and pilot clinical studies have reported that umbilical cord mesenchymal stem cells transplantation was a potential method to treat spinal cord injury, but its safety and efficacy remain controversial.

This study will conduct a multicenter, randomized, controlled trial for UC-MSC transplantation for the treatment of different phrases of SCI, including sub-acute, early stage, and late stage of chronic SCI. These three trials will investigate the safety and efficacy of intrathecal transplantation of UC-MSC in patients with SCI treatment. The study will be conducted at 3 hospitals in China, covering eastern, southern and western of Chinese mainland.

The primary outcome is the changes of motor and sensory assessment before and after intervention using American Spinal Injury Association (ASIA) Score Scale. Secondary outcomes will include International Association of Neural Restoration Spinal Cord Injury Functional Rating Scale (IANR-SCIRFS), electromyogram test, residual urine test and adverse events.

The enrolled participants will be followed up at baseline, 1, 3, 6 and 12 months after UC-MSC transplantation. Besides, the samples of serum and cerebrospinal fluid will be collected, before and after treatment, to explore the potential mechanism of UC-MSC transplantation for the treatment of SCI.

The results of this study will, for the first time, provide high level of evidence as to the relative safety and efficacy of UC-MSC transplantation for the treatment of spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Traumatic spinal cord injury
* ASIA Impairment Scale A-D
* Participants who understand and sign inform consent
* Duration of injury from 2 weeks to 2 months

Exclusion Criteria:

* Traumatic spinal cord injury with brain injury
* Non-traumatic spinal cord injury caused by spinal tumors, myelitis, demyelination, spinal vascular malformation, etc.
* with Ankylosing spondylitis
* with Malignant tumors
* with Neurodegenerative diseases, or any neuropathies
* with Hematologic diseases, or blood coagulation disorder
* with Hepatic dysfunction, renal dysfunction
* Ongoing or active infectious diseases
* Pregnancy, or lactation women
* Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent
* Not agree to take part in clinical trial or can't finish follow up
* Previous history of MSCs therapy
* Participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in American Spinal Injury Association (ASIA) Score Scale | baseline, 1 month, 3 months, 6 months and 12 months post-treatment
  Changes in motor and sensory scores assessed by the ASIA score scale (total score range from 0 to 324, higher values represent a better outcome)

SECONDARY OUTCOMES:
Changes in International Association of Neural Restoration Spinal Cord Injury Functional Rating Scale (IANR-SCIRFS) | Baseline, 1 month, 3 months, 6 months and 12 months post-treatment
  Changes in motor and sensory scores assessed by IANR-SCIRFS scale (total score range from 0 to 51, higher values represent a better outcome)
Changes in electromyogram test | Baseline, 6 months and 12 months post-treatment
  Changes in electromyogram test
Changes in residual urine | Baseline, 6 months and 12 months post-treatment
  Changes in residual urine measured by ultrasound test (volume of urine in mL, lower values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Limin Rong, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No